CLINICAL TRIAL: NCT02714959
Title: Effect of IL-2 in Refractory Autoimmune Encephalitis Patients: A Pilot Study
Brief Title: IL-2 in Refractory Autoimmune Encephalitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, Clinical Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510112713
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Encephalitis
MeSH Terms: conditions — Encephalitis | interventions — aldesleukin

ARMS (1):
- Proleukin (Experimental): Proleukin (subcutaneous injection) 1.5 MIU/day from day 1 to 5 at W1 3 MIU/day from day 1 to day 5 at W3, W6, and W9
  Interventions: Drug: Proleukin

INTERVENTIONS:
Drug: Proleukin

SUMMARY:
The purpose of this study is to determine whether low-dose IL-2 is effective in refractory autoimmune encephalitis.

DETAILED DESCRIPTION:
Autoimmune encephalitis is a recently recognized etiology of encephalitis which is mediated by various autoantibodies targeting neural cells or synapses. The responses to immunotherapy is generally good, considerable proportion of patients with autoimmune encephalitis have unfavorable clinical outcomes. Recently, depletion of regulatory T cell (Treg cell) is reported in variable autoimmune diseases and multiple studies have shown that low-dose interleukin-2(IL-2) specifically activates Treg cells to control autoimmunity and inflammation.

Protocol: This study is a single arm open-label study assessing clinical responses to the administration of low-dose IL-2 in autoimmune encephalitis patients who are refractory to first- and second-line immunotherapy.

Objective: To assess the efficacy of low-dose IL-2 in autoimmune encephalitis, resistant to first- and second- line immunotherapy.

Methods: This is a single arm open-label study. Each patients will receive four cycles of subcutaneous Proleukin (Interleukin-2, IL-2) (Week-1; 1.5 million IU (MIU)/d from Day-1 to Day-5, Week-3, -6, -9; 3MIU/d from Day-1 to Day-5) in the hospital. The patients will be followed up for 3 months (Week-21).

Primary outcome - clinical efficacy by modified Rankin Scale Secondary outcome - Immunologic follow-up of Treg cells before, during, and after IL-2 therapy, quality of life, cognitive function, side effect of low-dose IL-2

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical diagnosis of autoimmune encephalitis
* Positive for autoantibody (serum and or CSF) : NMDAR, anti-leucine-rich glioma inactivated-1(LGI-1), contactin-associated protein-like 2 (CASPR2), α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid receptor (AMPA) 1, AMPA2, GABAB-R, anti-Hu, -Yo, -Ri, -Ma2, -CV2/collapsing response mediator protein 5 (CRMP5), -amphiphysin, or glutamic acid decarboxylase (GAD)
* Refractory to first-line (high-dose steroid or intravenous immunoglobulin) and second line (rituximab or cyclophosphamide) immunotherapy
* Written informed consent form.

Exclusion Criteria:

* low hemoglobin <8.0 g/dL, absolute neutrophil count<1600/mm3, lymphocytes <600/mm3, platelets <140,000/mm3
* heart failure (≥ grade III NYHA), hepatic insufficiency (aspartate amino transferase >200 IU/L, amino alanine transferase, >200 IU/L), or lung failure
* Positive for HIV serology, active hepatitis B
* Significant abnormality in chest X-ray other than these linked to the diseases under investigation
* Infection
* Other progressive neurological degenerative disease.
* Poor venous access not allowing repeated blood tests
* pregnant or lactating women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Change of modified Rankin scale | Week 0,12

SECONDARY OUTCOMES:
The change of percentage of regulatory T (Treg) cells | Week 1, 3, 5, 9, 12, 21
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Week 1, 3, 5, 9, 12, 21
Quality of Life in Epilepsy Inventory (QOLIE)-31 | Week 21
  Quality of Life in Epilepsy Inventory (QOLIE)-31
Beck Depression Inventory (BDI) | Week 21
  Beck Depression Inventory (BDI)
Cognitive function | Week 21
  Mini-mental state examination (MMSE)

REFERENCES:
- [Background] Klatzmann D, Abbas AK. The promise of low-dose interleukin-2 therapy for autoimmune and inflammatory diseases. Nat Rev Immunol. 2015 May;15(5):283-94. doi: 10.1038/nri3823. Epub 2015 Apr 17. PMID 25882245
- [Background] Saadoun D, Rosenzwajg M, Joly F, Six A, Carrat F, Thibault V, Sene D, Cacoub P, Klatzmann D. Regulatory T-cell responses to low-dose interleukin-2 in HCV-induced vasculitis. N Engl J Med. 2011 Dec 1;365(22):2067-77. doi: 10.1056/NEJMoa1105143. PMID 22129253
- [Background] Hartemann A, Bensimon G, Payan CA, Jacqueminet S, Bourron O, Nicolas N, Fonfrede M, Rosenzwajg M, Bernard C, Klatzmann D. Low-dose interleukin 2 in patients with type 1 diabetes: a phase 1/2 randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2013 Dec;1(4):295-305. doi: 10.1016/S2213-8587(13)70113-X. Epub 2013 Oct 8. PMID 24622415
- [Background] Rosenzwajg M, Churlaud G, Mallone R, Six A, Derian N, Chaara W, Lorenzon R, Long SA, Buckner JH, Afonso G, Pham HP, Hartemann A, Yu A, Pugliese A, Malek TR, Klatzmann D. Low-dose interleukin-2 fosters a dose-dependent regulatory T cell tuned milieu in T1D patients. J Autoimmun. 2015 Apr;58:48-58. doi: 10.1016/j.jaut.2015.01.001. Epub 2015 Jan 26. PMID 25634360
- [Background] Castela E, Le Duff F, Butori C, Ticchioni M, Hofman P, Bahadoran P, Lacour JP, Passeron T. Effects of low-dose recombinant interleukin 2 to promote T-regulatory cells in alopecia areata. JAMA Dermatol. 2014 Jul;150(7):748-51. doi: 10.1001/jamadermatol.2014.504. PMID 24872229
- [Background] Humrich JY, von Spee-Mayer C, Siegert E, Alexander T, Hiepe F, Radbruch A, Burmester GR, Riemekasten G. Rapid induction of clinical remission by low-dose interleukin-2 in a patient with refractory SLE. Ann Rheum Dis. 2015 Apr;74(4):791-2. doi: 10.1136/annrheumdis-2014-206506. Epub 2015 Jan 21. No abstract available. PMID 25609413